CLINICAL TRIAL: NCT00204529
Title: Randomized, Multicenter, Open Label Study to Compare the Efficacy and Tolerability of Pegylated Interferon-alpha-2 (PEG-IFN) to 'Low-dose' Interferon-alpha-2a in Patients With Malignant Melanoma in Stages IIA (T3a) - IIIB (AJCC 2002)
Brief Title: Pegylated Interferon-alpha-2a in Patients With Malignant Melanoma Stage IIA-IIIB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Dermatologic Cooperative Oncology Group (Other)
Responsible Party: Principal Investigator, Thomas Eigentler, MD, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML17840
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Melanoma
Keywords: malignant melanoma; adjuvant therapy; Adjuvants, Immunologic
MeSH Terms: conditions — Melanoma | interventions — peginterferon alfa-2a; Interferon alpha-2

ARMS (2):
- PegIFN (Experimental): pegylated interferon-alpha-2a
  Interventions: Drug: pegylated interferon-alpha-2a
- IFN (Active Comparator): interferon-alpha-2a
  Interventions: Drug: interferon-alpha-2a

INTERVENTIONS:
Drug: pegylated interferon-alpha-2a
  Arms: PegIFN
Drug: interferon-alpha-2a
  Arms: IFN

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of adjuvant treatment with pegylated interferon-α-2a (PEG-IFN) vs. 'low dose' interferon-α-2a in patients with malignant melanoma in stage IIA (T3a) - IIIB.

A total of 880 will be randomized up to three months after first surgical management of their melanoma to either: PEG-IFN-α-2a or low-dose interferon-α-2a.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven cutaneous melanoma
* ≥ 18 years of age and < 75 years of age
* Have confirmed stage IIa (T3a), IIB, IIC, IIIA or IIIB (AJCC 2002) melanoma (lymph node staging either per sentinel node biopsy or elective lymph node dissection)
* Have a Karnofsky performance status of ≥ 80%
* Negative pregnancy test
* Start of therapy within three months after surgery
* Informed consent

Exclusion Criteria:

* Pregnant or lactating women
* Unwillingness or inability to employ an effective barrier method of birth control throughout the study and for up to 3 months after end of treatment in female or male patients
* Mucous membrane or ocular melanoma
* Any evidence of distant metastasis (CT-scan of brain, Chest X ray or CT, abdominal ultrasound or CT and ultrasound of regional lymph nodes at screening)
* Patients who have received chemotherapy or vaccines for melanoma
* Patients with tumor progression under a previous adjuvant interferon therapy or within three months after termination of interferon therapy (patients previously receiving adjuvant interferon therapy in another tumor stage without disease progression may be included)
* History of any other malignancy within the last ten years (except basal cell carcinoma or squamous cell carcinoma of the skin and carcinoma in situ of the cervix)
* Patients with severe cardiac disease (e.g. NYHA Functional Class III or IV, myocardial infarction within 6 months, ventricular tachyarrhythmias requiring ongoing treatment, unstable angina), severe liver disease or severe renal disease.
* ALAT or ASAT > 2 x ULN
* Bilirubin > 2 x ULN
* Creatinine > 2 x ULN
* Patients who have a history of depression or other psychiatric diseases requiring hospitalisation
* Patients with seizure disorders requiring anticonvulsant therapy
* Any of the following abnormal baseline hematologic/laboratory values:

  * Hb <10g/dl
  * WBC <3.0 x 109 /l
  * Platelets <100x109/l
  * Neutrophils < 1.5 x 109/l
* History or presence of autoimmune disease (i.e. autoimmune hepatitis, thyroid auto-immune dysfunction, systemic lupus erythematodes)
* Unwilling or unable to comply with the requirements of the protocol for the duration of the study
* Known infection with HBV, HCV, HIV
* Evidence of allergy or hypersensitivity against IFN or pegylated interferon
* Thyroid disease poorly controlled on prescribed medications
* Systemic corticosteroid therapy for any reason (>1 month)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 901 (Actual)
Dates: Start 2004-10 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Time to distant metastasis | From date of randomization until the date of first documented distant metastases or date of death from any cause, whichever came first, assessed up to 60 months

SECONDARY OUTCOMES:
Disease free survival | 5 years
Overall survival | 5 years
Quality of life | Measured at different visits (week 0, week 12, month 3, month 6)
Number and Grade of Adverse Events | Measured at every visit (week 4, week 8, week 12, month 3, month 6 and every 3 months during therapy)

CONTACTS AND LOCATIONS:
Overall Officials: Claus Garbe, MD, Principal Investigator — Skin Cancer Program, Department of Dermatology, University of Tübingen, Liebermeisterstr. 20, 72076 Tübingen, Germany; Hubert Pehamberger, MD, Principal Investigator — Department of Dermatology, University Hospital Vienna, Währinger Gürtel 18-20, 1090 Vienna, Austria
Locations (1):
- Arbeitsgemeinschaft Dermatologische Onkologie, Skin Cancer Program, Department of Dermatology, University of Tübingen, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Eigentler TK, Gutzmer R, Hauschild A, Heinzerling L, Schadendorf D, Nashan D, Holzle E, Kiecker F, Becker J, Sunderkotter C, Moll I, Richtig E, Ponitzsch I, Pehamberger H, Kaufmann R, Pfohler C, Vogt T, Berking C, Praxmarer M, Garbe C; Dermatologic Cooperative Oncology Group (DeCOG). Adjuvant treatment with pegylated interferon alpha-2a versus low-dose interferon alpha-2a in patients with high-risk melanoma: a randomized phase III DeCOG trial. Ann Oncol. 2016 Aug;27(8):1625-32. doi: 10.1093/annonc/mdw225. Epub 2016 Jun 10. PMID 27287206
- See also: Synopsis of study protocol — http://www.hauttumorzentrum.de